CLINICAL TRIAL: NCT04515836
Title: Phase II Trial of Olaparib in Homologous Recombination Deficient (HRD) Malignant Mesothelioma
Brief Title: Olaparib in Patients With HRD Malignant Mesothelioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-0117
Record Dates: First submitted 2020-07-18; First posted 2020-08-17 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Mesothelioma; Homologous Recombination Deficiency
Keywords: mesothelioma, lung cancer, malignant mesothelioma
MeSH Terms: conditions — Mesothelioma; Lung Neoplasms; Mesothelioma, Malignant | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Olaparib will be given orally to patients in 28-day cycles. Patients will attend the clinic on days 1 (first day of treatment) and 15 of the first cycle following the beginning of study treatment and then every 4 weeks (day 1 of every cycle) until discontinuation of treatment.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib is a chemotherapy drug (packaged as a pill) that can be taken by mouth, twice daily.
  Other Names: Lynparza

SUMMARY:
In this study, researchers will give olaparib (a drug) to mesothelioma patients who have specific changes in their DNA (known as gene mutations). Researchers will give this drug to each patient on the study to find out if it will help the patient's tumor shrink or stop growing.

ELIGIBILITY:
Inclusion Criteria:

* Must have a medical diagnosis of malignant mesothelioma that has been confirmed by a physician.
* Participant must be able to sign a consent form stating that they choose (of their own free will) to participate in the study and agree to follow the study requirements and restrictions that are listed in the consent form.
* Must be willing to sign and date consent form before any mandatory study-specific procedures, sample collecting and tests.
* Willing to experience genetic testing to determine study eligibility. Must be willing to genetically test tumor and normal body cells.
* Before participating in the treatment phase of this study, participants must be willing to give their own consent (agreement) to have their samples collected for genetic and biomarker research.
* Age 18 or older.
* Participant must show evidence of specific DNA changes/genetic mutations defined as follows: A) BAP1 loss (the loss of a protein called ubiquitin carboxyl-terminal hydrolase) verified by physicians at the University of Chicago using sampling tests AND/OR B) A mutation (abnormal change) in the participant's germ cells (reproductive cells) or somatic cells (non-reproductive cells) that disrupts protein function in at least one of the patient's genes.
* Prior treatment with cisplatin or carboplatin is required.
* Patients must have platinum-sensitive disease (cancer that responds to treatments with anticancer drugs containing metal platinum). For eligibility in this study, platinum-sensitive disease will be defined as no disease progression while on a platinum agent (chemotherapy drug) or for at least 3 months after completing treatment with a platinum agent.
* Patients must have normal organ and bone marrow function measured within 28 days prior to receiving study treatment. Normal bone marrow and organ function will be assessed using specific lab tests/ criteria set by the study's lead physician.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients must have a life expectancy of 16 weeks or more.
* Must have a tumor that can be measured according to criteria set by the modified Response Evaluation Criteria in Solid Tumors (RECIST) standards for pleural mesothelioma and RECIST 1.1 for peritoneal and tunica vaginalis mesothelioma. Patients in the study must have at least one area of damaged tissue (a lesion) that has not received previous radiation treatment. This damaged tissue must be accurately measured at the beginning of the study as greater than or equal to 10 mm in the longest diameter (except lymph nodes which must have short axis greater than or equal to 15 mm). The patient's tumor would be measured using computed tomography (CT), which is suitable for accurate repeated measurements.
* Both male and female patients can participate in this study.
* If a woman is of childbearing potential and wishes to participate in the study, she most show evidence that she is not pregnant using a negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.
* Women who are postmenopausal and wish to participate in the study, must also show evidence of postmenopausal status. Postmenopausal status will be defined as: 1) A woman who does not experience menstruation (known as amenorrhea) for 1 year or more following the end of hormonal treatments. 2) Women who have reproductive/hormone levels in the post-menopausal range for women under 50 as confirmed by medical tests; 3) Radiation-induced oophorectomy (removal of one or more ovaries) with last menses greater than 1 year ago; 4) Menopause caused by chemotherapy with greater than 1 year since last menses 5) Surgical sterilization (bilateral oophorectomy or hysterectomy).
* Male patients must use a condom during treatment and for 3 months after the last dose of study drug (olaparib) when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.
* NOTE 1: Tests to confirm the eligibility of participants who have the above mutations (altered germ or somatic cells) will take place at a germline or tumor sequencing lab that is certified under the Clinical Laboratory Improvement Amendments (CLIA). Eligibility of study participants will be confirmed once the physical leading this study receives the official mutation report from the lab and confirms that the participant's identified mutation fits the definition outlined above. All other patients must consent to tumor and normal sample sequencing as described in study procedures below during the prescreening phase to determine eligibility.
* NOTE 2: Rare exceptions of participants who may have conflicting evidence regarding protein function will be interpreted on an individual basis by the physician leading the study.

Exclusion criteria:

Medical conditions:

* Any evidence of uncontrollable illness that the physician leading this study deems undesirable for the patient to participate in the trial.
* Other malignancy (tumor/cancer) unless it has been treated with no evidence of disease for 3 or more years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.
* Patients with BAP1 tumor predisposition syndrome will be included in the trial. These patients may be eligible if they have a history of syndrome-related cancers, provided they completed their surgery and chemotherapy more than three years prior to registration, and the patient remains free of disease that continues to re-occur or spread to other parts of the body.
* Patients with cancer that does not respond to platinum chemotherapy drugs (known as platinum-resistant disease), defined as disease progression during or within 3 months of receiving chemotherapy.
* Resting electrocardiogram (ECG) that shows the patient has uncontrolled, potentially reversible cardiac conditions or patients with congenital long QT syndrome (a heart rhythm condition that can cause fast, chaotic heartbeats), as judged by the study's lead physician.
* Persistent toxicities (greater than the Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
* Patients with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with findings suggestive of MDS/AML.
* Patients with cancer cells that have moved from one part of their body to the brain (brain metastases) causing the patient to show symptoms/signs of more serious illness. A scan to confirm the absence of cancerous cells in the brain is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
* Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-cancerous systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Patients unable to swallow oral medications and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients who have a compromised immune system, e.g., patients who have tested positive for human immunodeficiency virus (HIV).
* Patients with known active hepatitis (i.e. Hepatitis B or C) confirmed by medical tests; patients with a past or resolved Hepatitis B infection are eligible. Patients positive for hepatitis C virus are eligible only if samples of the patient's DNA tests negative for hepatitis C, according to genetic tests (using polymerase chain reaction).

Prior/concomitant therapy (medications/treatments that may conflict with the study drug, olaparib):

* Any previous treatment with a type of drug/substance called a PARP inhibitor (which stands for poly-ADP ribose polymerase inhibitor), including olaparib.
* Receipt of any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment.
* Patients who are using strong cancer drugs called CYP3A inhibitors (also called Cytochrome P-450) for treatment (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). Any treatment previously taken by the patient must be washed out of the patient's system 2 weeks before taking olaparib in this study.
* Patients who are using known strong CYP3A inducers (drugs for cancer patients including phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). Any patients taking enzalutamide must have the drug washed out of their system 5 weeks before stating olaparib in this study; patients taking phenobarbital and other agents must have the drug washed out of their system 3 weeks before taking olaparib in this study.
* Major surgery within 2 weeks of starting study treatment; patients must have recovered from any effects of any major surgery.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).

Prior/concurrent clinical study experience:

* Participation in another clinical study where the patient received a study drug in the last month before starting this study.
* Patients with a known hypersensitivity to olaparib or any of the ingredients in the product.

Other exclusions:

* Involvement in the planning and/or conduct of the study.
* The lead study physician deciding that the patient should not participate in the study if the patient is unlikely to follow study procedures, restrictions and requirements.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2028-04-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate of Patients to Olaparib | Two years.
  To determine the percentage of patients with mesothelioma tumors (containing certain gene/cell mutations) that shrink or stop growing as a response to olaparib.

SECONDARY OUTCOMES:
Overall Survival of Patients Taking Olaparib | Three years.
  To determine the length of time patients on the study are still alive after taking olaparib.
Progression-Free Survival of Patients Taking Olaparib | Two years.
  To determine the length of time patients taking olaparib can live with mesothelioma without their cancer getting worse.
Frequency of Treatment-Related Side Effects/ Adverse Events | Two years.
  To determine the frequency of treatment-related side effects/ adverse events reported among study participants. These side effects will be assessed by attribution (source), type and grade. Adverse events/side effects will be graded using the NCI Common Terminology Criteria for Adverse Events (Version 5).

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L Kindler, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States